CLINICAL TRIAL: NCT04404413
Title: Effect of High-Intensity Interval Training and Intermittent Fasting on Body Composition and Physical Performance in Active Women
Brief Title: High-Intensity Interval Training and Intermittent Fasting on Body Composition and Physical Performance in Active Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alicante (Other)
Collaborators: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Prof. Dr. Alejandro Martínez-Rodríguez, Assistant Professor, University of Alicante
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CE061811
Record Dates: First submitted 2020-05-19; First posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Body Composition; Physical Performance; Intermittent Fasting
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PARTICIPANTS (Experimental): A single-group crossover design was used to compare the effects of 2x8 weeks of high-intensity interval training without (HIIT) or with (HIIT+IF) intermittent fasting caloric restriction (20% reduction in weekly energy intake) on body composition and performance. There were two weeks in the middle of both phases in which they did not carry out programmed activity, in order not to alter the experimental phase.
  Interventions: Behavioral: Intensity interval training (HIIT); Behavioral: Intensity interval training (HIIT) + intermittent fasting

INTERVENTIONS:
Behavioral: Intensity interval training (HIIT) — 2x8 weeks of high-intensity interval training (HIIT)
Behavioral: Intensity interval training (HIIT) + intermittent fasting — 2x8 high-intensity interval training with (HIIT+IF) intermittent fasting caloric restriction (20% reduction in weekly energy intake).

SUMMARY:
The objective of this study is to compare the body composition and physical performance effects of HIIT, with or without intermittent fasting intervention in active women. Fourteen active normal weight women aged 18-35 participated in the study. The effects of 2x8 weeks without (HIIT) or with (HIIT+IF) intermittent fasting caloric restriction (20% reduction in weekly energy intake) on body composition and performance (Hand-grip strength, Counter movement jump, Wingate Anaerobic 30 s Cycling Test), were compared. There were two weeks in between both phases when they did not perform the scheduled activity, so as not to alter the experimental phase.

ELIGIBILITY:
Inclusion Criteria:

1. No muscular, ligamentous, bone, nerve or joint pathology incompatible with the training program.
2. Not to present cardiovascular or cardiorespiratory problems.
3. Physically active in the last 5 years, according to the American College of Sports Medicine (ACSM) definition.

Exclusion Criteria:

1. Following pharmacological treatment or supplement.
2. Performing other sports activities that may influence the study results during their participation in the study.
3. Not following training or diet program guidelines or attending scheduled training sessions.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Hand-grip strength | 16 weeks
  Hand-grip strength test was performed as an indicator of overall strength.
Counter movement jump (CMJ) | 16 weeks
  In the CMJ test, the participants performed a maximum vertical jump starting from a standing position with arm swing not allowed.
Wingate Anaerobic 30 s Cycling Test | 16 weeks
  Wingate Anaerobic 30 s Cycling Test with a validated cycloergometer (Monark 894E, Vansbro, Sweden).
Fat mass | 16 weeks
  Body composition masses were estimated using validated equations. Carter's equation was used to estimate fat mass.
Muscle mass | 16 weeks
  Body composition masses were estimated using validated equations. Lee's equation to estimate muscle mass.
Residual mass | 16 weeks
  Body composition masses were estimated using validated equations. Residual mass was obtained from the difference between fat mass and muscle mass.
Body Mass | 16 weeks
  It was performed using a digital scale with 0,1kg accuracy (Tanita BC-545, Tokyo, Japan).

CONTACTS AND LOCATIONS:
Locations (1):
- Alejandro Martínez Rodriguez, San Vicent del Raspeig, Alicante, Spain